CLINICAL TRIAL: NCT06226584
Title: Therapeutic Effects of Multiple-strain Probiotics for Children With ADHD Based on Assessment of Standardized Attention Tests and Quantitative Electroencephalogram: a Single Arm Pilot Study
Brief Title: Multi-strain Probiotics for ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tsyr-Huey Mental Hospital (Other)
Responsible Party: Principal Investigator, Cheng Yu-Shian, Psychiatrist, Tsyr-Huey Mental Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MultiProbioADHD
Record Dates: First submitted 2024-01-13; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Attention Deficit and Hyperactivity Disorders
Keywords: ADHD; probiotics; quantitative electroencephalogram
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- multiple-strain probiotics (Experimental)
  Interventions: Dietary Supplement: multiple-strain probiotics

INTERVENTIONS:
Dietary Supplement: multiple-strain probiotics — Juice HA capsule which contains more than one strain of probiotics

SUMMARY:
Probiotics are widely used as supplement for various neurodevelopmental disorders. The mechanism of their therapeutic potential lies in the "gut-brain axis", a two-way communication pathway through the neuroendocrine system. In the past, there have been many experiments to study the possible efficacy of probiotics in patients with ADHD. Although some studies have shown that probiotics can improve ADHD symptoms, most studies have used behavioral rating scales to evaluate. As a result, it is susceptible to informant bias. Standardized attentional tests and quantitative electroencephalogram (qEEG) can provide more objective data and detect possible changes in brain networks. Such changes may precede behavioral phenotypes. Therefore, the purpose of this study is mainly to detect the therapeutic effect of multiple strains of probiotics in patients with attention deficit hyperactivity disorder by using standardized attention tests and quantified brain waves (qEEG).

ELIGIBILITY:
Inclusion Criteria:

A patient is eligible for the study if all of the followings apply:

1. 8-11 children diagnosed with ADHD by board certified pediatric psychiatrist according to DSM-5 (assessment tool using SNAP criteria, at least 6/9 symptoms of inattention and/or hyperactivity/impulsivity (≧2/3 on each severity scale) on parents' and teachers' observation)
2. On stable psychotropic mediations (i.e. no change in dose of methylphenidate or antipsychotics) for past 8 weeks

Exclusion Criteria:

Any patient meeting any of the exclusion criteria will be excluded from study participation:

1. Patients with major mental or neurological diseases such as intellectual disability, autism group disorders, schizophrenia, severe depression, bipolar disorder, epilepsy, brain injury, etc.
2. Those who have serious gastrointestinal diseases, physiological diseases or genetic diseases.
3. Have used antibiotics or edible probiotic-related products (including drops, tablets, capsules, bacterial powder) in the past month.
4. Participated in other clinical research in the past month.
5. Vegetarians or those currently undergoing special diet therapy.
6. Evaluation by the pediatric psychiatrist not suitable for entering the test

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
The Swanson, Nolan and Pelham Chinese (SNAP) rating scales | every one month for 3 months
  for behavioral symptoms of ADHD, the minimum and maximum values (0-78), higher scores mean a worse outcome
Conners' Continuous Performance Test 3rd Edition | pre- and post-intervention (3 months)
  a task-oriented computerised assessment of attention-related problems in individuals aged 8 years and older
quantitative electroencephalogram | pre- and post-intervention (3 months)
  measurement of brain wave patterns and coherence

SECONDARY OUTCOMES:
adverse events | every one month for 3 months
  any adverse events occurred during study

CONTACTS AND LOCATIONS:
Overall Officials: YU-SHIAN CHENG, MDPhD, Principal Investigator — Tsyr-Huey Mental Hospital
Locations (1):
- Tsyr-HueyMentalHospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No